CLINICAL TRIAL: NCT03137732
Title: Surgical Placement Versus Anaesthetic Placement of Rectus Sheath Catheter for Pain Relief Following Major Abdominal Surgery (SPARC). A Single Centre Randomised Controlled Trial
Brief Title: Surgical Versus Anaesthetic Placement of Rectus Sheath Catheters
Acronym: SPARC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Countess of Chester NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dale Vimalachandran, Consultant Colorectal Surgeon, Countess of Chester NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Surg 058/17
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Last update posted 2017-05-03 (Actual); Status verified 2017-04

CONDITIONS: Pain, Postoperative; Wound; Abdomen; Incision
MeSH Terms: conditions — Pain, Postoperative; Abdominal Injuries; Surgical Wound

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to the intervention that they are randomized to intraoperatively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgeon-inserted (Active Comparator): Rectus sheath catheter will be inserted under direct vision / palpation of the space at the end of the operation.
  Interventions: Device: Rectus Sheath Catheter
- Anaesthetist-inserted (Active Comparator): Rectus sheath catheter will be inserted under ultrasound guidance by the anaethetist.
  Interventions: Device: Rectus Sheath Catheter

INTERVENTIONS:
Device: Rectus Sheath Catheter — Insertion of rectus sheath catheter via either method

SUMMARY:
This is a single centred randomized controlled trial comparing surgeon versus anaesthetist inserted rectus sheath catheters for management of analgesia post major abdominal surgery.

DETAILED DESCRIPTION:
Background and study aims Pain management post laparotomy (abdominal surgery) can be difficult and in our trust we are increasingly using rectus sheath catheters (RSCs).This is achieved by placing catheters, done by either by the surgeon or anaesthetist into the potential space between the rectus muscle and the posterior rectus sheath. Two catheters are placed, one on either side of the mid-line wound. Local anaesthetic is then infused through the catheters for up to 3 days post-operatively. This provides analgesia to the central abdominal wall in the region of the T7-T11 dermatomes. It only provides analgesia for somatic pain, not visceral pain and hence needs to be used in addition to a multi-modal analgesic regime usually including a patient controlled analgesia device (PCA) containing either morphine or oxycodone. Advantages of a RSC infusion over an epidural include that it can be used in patients with coagulopathy or systemic infection and can be safely performed asleep. It is also less labour intensive to manage on the ward and does not carry the same risks of hypotension and excessive fluid administration that are associated with an epidural.

There is randomised controlled trial evidence that RSC infusions in addition to PCA provide superior analgesia when compared to PCA alone in surgery performed through a midline incision. There is also a randomised controlled trial in progress that is comparing analgesic quality of epidural infusions to RSC with PCA. In most published literature to date, RSC are inserted by the anaesthetist using ultrasound to aid placement. In our hospital, some RSC are inserted by anaesthetists although the majority are performed by surgeons at the end of an operation. This is because we believe that this technique is less time consuming and both insertion techniques result in equivalent analgesia.

The primary aim endpoint of this study is to determine any difference in insertion time for rectus sheath catheters between those inserted by surgeons and those inserted by anaesthetists. Observationally in our hospital, there is no difference in quality of analgesia provided by the two insertion techniques. However, surgical insertion of RSC causes less disruption of an operation as the patient already has their abdomen draped with sterilised skin as part of their surgical procedure. Also, surgical insertion of RSC with an open abdomen is potentially easier than ultrasound guided insertion by an anaesthetist before an operation.

Who can participate? Any adults undergoing emergency or elective laparotomy (major abdominal surgery.) What does the study involve? All participants will receive rectus sheath catheters but will be randomly allocated to each group. Following the surgery, participants will have to answer questions about their pain on 3 consecutive days.

What are the possible benefits and risks of participating? There are no specific benefits to patients and the risks are the same if they were in the trial or not as it is routine in our hospital to use rectus sheath catheters as a means of analgesia post laparotomy. These risks include bleeding, dislodgement of catheter and failure of catheter and are low risk.

Where is the study run from? This a single centre study at the Countess of Chester Hospital in the United Kingdom.

When is study starting and how long is it expected to run for? We anticipate recruiting patient from June 2017 for 6 months. How long will the trial be recruiting participants for? No funding is required as all data collection will be carried out by doctors working in the departments but the study is being supported and supervised by the Hospital's Research and Development department.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Able to provide informed consent
* Undergoing elective, open colorectal surgery or emergency laparotomy via a midline incision extending above the umbilicus
* Weight of 50kg or over to standardise the analgesia given.

Exclusion Criteria:

* Weight of less than 50kg
* Patients unable to consent
* Age under 18 years
* Inability to insert RSC - local infection or severe coagulopathy
* Allergy to local anaesthetic
* Chronic pre-operative use of strong opioids or gabapentins and or chronic pain syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Time taken to insert rectus sheath catheters | under 15 minutes
  This will be recorded in theatre on a stopwatch and recorded.

SECONDARY OUTCOMES:
Pain scores | 4 days
  Patients will be asked to score their pain in recovery and on days 0,1,2,3 post operatively. This will be graded using a Numeric Pain Rating Scale.
Peri-operative analgesic use | 4 days
  Analgesic use intra-operatively and post-operatively for 3 days. This will include strong opioids, paracetamol, NSAIDs, codeine, ketamine, IV lignocaine, tramadol, clonidine and PCA usage post-operatively.
Catheter issues | 4 days
  This includes haemorrhage, dislodgement, blockage
Duration of catheter use | 4 days
TIme to diet and mobilisation | likely 1-3 days
Time to discharge | approximately 7 days

IPD SHARING:
Plan to Share IPD: Undecided